CLINICAL TRIAL: NCT03466528
Title: A Prospective Randomised Controlled Trial of the Effect of Magnesium Sulphate Administration on Red Cell Transketolase Activity in Alcohol Dependent Patients at Risk of Wernicke Korsakoff Syndrome Treated With Thiamine
Brief Title: Alcohol: Thiamine and or Magnesium 1
Acronym: AToM1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Glasgow Royal Infirmary (Other)
Responsible Party: Principal Investigator, Dr. Donogh Maguire, Emergency Medicine Consultant, Glasgow Royal Infirmary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN16ME174; 201773 (Other: IRAS)
Record Dates: First submitted 2018-02-13; First posted 2018-03-15 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Alcohol Withdrawal; Lactic Acidosis; Vitamin B1 Deficiency; Magnesium Deficiency; Wernicke Encephalopathy
MeSH Terms: conditions — Acidosis, Lactic; Beriberi; Magnesium Deficiency; Wernicke Encephalopathy | interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: This is a 3- arm randomised, open label, controlled study in a cohort of alcoholic patients admitted through A&E. Patients will be randomised to concurrent infusion of one of the following:
  * Arm 1: IV thiamine
  * Arm 2: IV magnesium sulphate followed by delayed IV thiamine
  * Arm 3: IV thiamine and IV magnesium sulphate Thiamine will be administered as IV Pabrinex, a compound preparation which also contains B vitamins and vitamin C. Administration of IV Pabrinex is standard care in this patient group and magnesium sulphate is routinely co-administered at Glasgow Royal Infirmary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard treatment - Pabrinex alone (Active Comparator): Pabrinex alone
  Interventions: Drug: Pabrinex
- Pabrinex + magnesium sulphate (Active Comparator): standard treatment and magnesium sulphate
  Interventions: Drug: Magnesium Sulfate; Drug: Pabrinex
- Magnesium sulphate alone (Experimental): This group receives the study intervention and delayed Pabrinex
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Intravenous (Magnesium Sulphate) MgSO4 2 grams IV over 20 minutes
  Other Names: MgSO4
  Arms: Magnesium sulphate alone; Pabrinex + magnesium sulphate
Drug: Pabrinex — standard treatment
  Other Names: comercial form of thiamine and B vitamin preparation
  Arms: Pabrinex + magnesium sulphate; Standard treatment - Pabrinex alone

SUMMARY:
Patients who suffer Alcohol Use Disorder (AUD) have a 30-80% incidence of thiamine deficiency causing Wernicke's Encephalopathy (WE).

Intravenous (IV) thiamine replacement is standard practice in the treatment of alcoholic patients presenting to the Accident & Emergency (A&E) department, however routine co-supplementation with magnesium (administered IV as magnesium sulphate ), which is required as a co-factor for thiamine in some metabolic processes, e. g. on the activity of the enzyme transketolase in red blood cells, is not routine practice in the treatment of these patients. Without correction of concomitant magnesium deficiency there may be impaired utilisation of thiamine resulting in a failure to treat WE.

This study is designed to determine if administration of magnesium to AUD patients affects red cell transketolasae and serum lactate concentrations by itself, or only acts to increase the effect of thiamine on the activity of this enzyme.

DETAILED DESCRIPTION:
This is a 3- arm randomised, open label, controlled study in a cohort of alcoholic patients admitted through A&E. Patients will be randomised to concurrent infusion of one of the following:

* Arm 1: IV thiamine
* Arm 2: IV magnesium sulphate followed by delayed IV thiamine
* Arm 3: IV thiamine and IV magnesium sulphate Thiamine will be administered as IV Pabrinex, a compound preparation which also contains B vitamins and vitamin C. Administration of IV Pabrinex is standard care in this patient group and magnesium sulphate is routinely co-administered at Glasgow Royal Infirmary.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male or non-pregnant or breastfeeding females ≥18 years of age For women of child-bearing potential a negative pregnancy test will be required prior to treatment.

(Women of non-childbearing potential are defined as those defined as women who are post-menopausal or permanently sterilised (e.g. hysterectomy, tubal occlusion, bilateral salpingectomy).

• Chronic alcohol dependence as confirmed by

* FAST questionnaire
* GMAWS scale

Exclusion Criteria:

* Unable to give consent
* Less than 18 years of age
* Chronic renal or hepatic failure/hepatic encephalopathy (investigator assessment as documented in past medical history i.e. Clinical Portal.)
* Known hypersensitivity or previous allergy to any of the active substances in either trial medication, or to excipients
* Severe concurrent medical condition that would prevent participation in study procedures (e.g. myasthenia gravis, clinically significant cardiac disease, or cardiac failure with severe pulmonary oedema)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Change in Erythrocyte transketolase activity | 0 and 2 hours
  this is a biochemical marker of thiamine activity measured in units per gram of haemoglobin
Change in serum lactate | 0 and 2 hours
  Biochemical marker of metabolic dysfunction (expressed as mmol/L)
Change in rate of resolution of alcohol withdrawal syndrome | days
  time

SECONDARY OUTCOMES:
lactate dehydrogenase | 0 and 2 hours
  biochemical (expressed in mmol/L)
pre and post magnesium | 0 and 2 hours
  biochemical (expressed in mmol/L)
pre and post red cell thiamine | 0 and 2 hours
  biochemical
establish baseline micronutrient status of patients with alcohol withdrawal syndrome | o and 2 hours
  biochemical

CONTACTS AND LOCATIONS:
Overall Officials: Donogh Maguire, MB BCh, Principal Investigator — NHS GGC
Locations (1):
- Glasgow Royal Infirmary, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maguire D, Burns A, Talwar D, Catchpole A, Stefanowicz F, Ross DP, Galloway P, Ireland A, Robson G, Adamson M, Orr L, Kerr JL, Roussis X, Colgan E, Forrest E, Young D, McMillan DC. Randomised trial of intravenous thiamine and/or magnesium sulphate administration on erythrocyte transketolase activity, lactate concentrations and alcohol withdrawal scores. Sci Rep. 2022 Apr 28;12(1):6941. doi: 10.1038/s41598-022-10970-x. PMID 35484175

DOCUMENTS (2):
  • Informed Consent Form (2016-09-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT03466528/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/28/NCT03466528/Prot_SAP_001.pdf